CLINICAL TRIAL: NCT03429413
Title: Maximizing HPV Vaccination: Real-time Reminders, Guidance, and Recommendations - Part 4: Feasibility Trial
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Patient-Centered Outcomes Research Institute (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: IRB201701537 -N; R21CA202011 (NIH); OCR19940 (Other: UF OnCore)
Record Dates: First submitted 2018-02-05; First posted 2018-02-12 (Actual); Last update posted 2025-08-17 (Actual); Status verified 2025-08

CONDITIONS: Human Papillomavirus (HPV) Vaccines
Keywords: Health Information Technology (HIT)
MeSH Terms: conditions — Papillomavirus Infections

STUDY DESIGN:
Intervention Model Description: Clinics are randomly assigned to use the intervention app or not. A 5th clinic, will use the app, but has not been involved in the app development.
Who Masked: Outcomes Assessor
Masking Description: The statistical team is blinded to the clinic assignment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Parents (Active Comparator): Parents of 11-12 year old children who visit participating interventional clinics during study period.
  Interventions: Behavioral: Protect Me 4 Application + External Quality Improvement Support; Behavioral: Protect Me 4 Application Alone
- Health Care Provider (Active Comparator): Health care providers and clinic staff for 11-12 year old patients at 4 participating pediatric clinics.
  Interventions: Behavioral: Protect Me 4 Application + External Quality Improvement Support; Behavioral: Protect Me 4 Application Alone
- Adolescents at Intervention clinics (No Intervention): Adolescents between 11-12 years of age. Adolescent vaccination data is used in the study, adolescents will assent to participate. The parents, however, use the HIT system.
- Adolescents at Control Clinic (No Intervention): Parents of 11-12 year old children who visit participating control clinics during study period.
- Health Care Provider at Control Clinic (No Intervention): Health care providers and clinic staff for 11-12 year old patients at 3 participating pediatric control clinics.

INTERVENTIONS:
Behavioral: Protect Me 4 Application + External Quality Improvement Support — Participants will be asked to interact with the Protect Me 4 application, using an iPad tablet. During the implementation period (months 4-6), intervention clinics will receive the Protect Me 4 app and External Quality Improvement Support (practice facilitation and external and internal provider peer opinion leaders and provider incentives). Providers from intervention clinics will complete audit and feedback reports to assess HPV vaccination rates with the assistance of the practice facilitator. Providers at the intervention clinic will complete a pre-intervention survey to obtain background information (demographics, approximate HPV vaccination rates, comfort with the use of technology etc.)
  Arms: Health Care Provider; Parents
Behavioral: Protect Me 4 Application Alone — During the maintenance period (months 7-9), intervention clinics will receive Protect Me 4 without external support (practice facilitation and external provider peer opinion leaders). Providers from intervention clinics will complete audit and feedback reports to assess HPV vaccination rates without the assistance of the practice facilitator. Providers at the intervention clinic will complete a post-intervention survey to gain provider feedback regarding the feasibility of Protect Me 4 and changes in perceptions regarding the use of technology.
  Other Names: Enhanced HIT System Intervention
  Arms: Health Care Provider; Parents

SUMMARY:
Human papillomavirus (HPV) vaccines have potential to prevent an average of 26,900 cancer cases each year in the United States, but vaccine coverage rates remain low. The study team has developed an electronic application (app), Protect Me 4, to help parents and providers assess and have more productive conversations about needed vaccines.

The specific aims of this study are to: (1) evaluate the feasibility of implementing Protect Me 4, and (2) estimate preliminary efficacy of Protect Me 4 to increase HPV vaccine initiation (receipt of first dose).

DETAILED DESCRIPTION:
Human papillomavirus (HPV) vaccines have potential to prevent an average of 26,900 cancer cases each year in the United States, but vaccine coverage rates remain low. The study team has developed a health information technology (HIT) electronic application (app), Protect Me 4, to help parents and providers assess and have more productive conversations about needed vaccines.

In past studies, Protect Me 4 users have demonstrated three times higher chances of initiating the HPV vaccine. Despite this promise, Protect Me 4 system implementation suffered from very low reach within clinics. In this phase of the project, the investigators will assess the feasibility of implementing Protect Me 4 in community clinics, as well as test vaccination rate data collection strategies and estimate the preliminary efficacy of Protect Me 4 to increase HPV vaccine initiation. Seven clinics will participate in the study, and three will be randomly assigned the use of Protect Me 4. Three of the clinics will act as controls and will not receive Protect Me 4. The final clinic will receive the intervention (but has not participated in any of the intervention development. This clinic will s as a demonstration clinic for the subsequent R01.

For evaluation, vaccination records will be grouped in three-month periods [initial (months 1-3), implementation (months 4-6) and maintenance (months 7-9)] from Medicaid and CHIP (Children's Health Insurance Program) claims and Florida Immunization Registry data. During the implementation period (months 4-6), intervention clinics will receive the Protect Me 4 app and External Quality Improvement Support (practice facilitation and external and internal provider peer opinion leaders and provider incentives). During the maintenance period (months 7-9), intervention clinics will receive Protect Me 4 without external support (practice facilitation and external provider peer opinion leaders).

To evaluate effectiveness at the individual-level, the study team will compare vaccination rates between eligible adolescents who visited intervention and control clinics across the three time periods.

ELIGIBILITY:
Inclusion Criteria:

* Must be parent of an adolescent aged 11-12 years old.
* Providers working with age appropriate for study adolescents at the intervention clinics
* Adolescents/Parents/Providers willing to consent to participation
* Adolescents/Parents that can read and speak English

Exclusion Criteria:

* Adolescents out of the age range for participation
* Adolescents/Parents/Providers unwilling to consent to participation
* Adolescents/Parents that can NOT read and speak English

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1296 (Estimated)
Dates: Start 2026-09-15 (Estimated); Primary Completion 2027-09-15 (Estimated); Study Completion 2027-09-15 (Estimated)

PRIMARY OUTCOMES:
Reach - Feasibility | After month 9
  Goal will be to have 80% of the parents of 11-12 year olds offered the Protect Me 4 app.
Adoption - Feasibility | After month 9
  Goal will be to have 70% of parents complete the Protect Me 4 app for each provider. App will be considered feasible of 80% or more of providers use the app during the study.
Provider-level Implementation - Feasibility | After month 9
  Goal will be to have providers report using the discussion tips approximately half the time they are provided and offering HPV vaccine 75% of the time it is due. App will be considered feasible if providers view shot lists for 60% of their patients with screens indicating that shots are due. Will aim for providers to look at specific hesitations reported by parents 60% of the time they login to the app and hesitations are reported.
Parent-level Implementation - Feasibility | After month 9
  Goal will be to have 95% of people who start the app successfully enter the app and 80% agree to participate (consent and assent.)
Maintenance - Feasibility | Months 7-9
  During months 7-9, the study team will assess clinic and provider maintenance of use of the Protect Me 4 app
Acceptability - Feasibility | Month 6, Month 9
  At both the end of the implementation and the maintenance period, providers will complete the Post Intervention Survey.

SECONDARY OUTCOMES:
Data Collection Strategy | After month 9
  Analysis of de-identified participant datasets linked to clinic records, HIT participation date, and vaccinations from the Florida Medicaid and CHIP claims or the Florida Immunization Registry data.
Efficacy Measurements | After month 9
  Determination of HPV vaccine initiation using Current Procedural Terminology (CPT) and Current Vaccine Administered (CVX) codes

CONTACTS AND LOCATIONS:
Overall Officials: Stephanie Staras, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States